CLINICAL TRIAL: NCT04006210
Title: A Multicenter, Randomized, Active-controlled, Double-blind, Double-dummy, Parallel-group Clinical Trial, Investigating the Efficacy, Safety, and Tolerability of Continuous Subcutaneous ND0612 Infusion in Comparison to Oral IR-LD/CD in Subjects With Parkinson's Disease Experiencing Motor Fluctuations (BouNDless)
Brief Title: Efficacy, Safety and Tolerability Study of ND0612 vs. Oral Immediate Release Levodopa/Carbidopa (IR-LD/CD) in Subjects With Parkinson's Disease Experiencing Motor Fluctuations
Acronym: BouNDless
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND0612-317
Record Dates: First submitted 2019-06-30; First posted 2019-07-05 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Oral IR-LD/CD Adjustment Period - Run-in 1 (1 arm) followed by ND0612 Conversion Period - Run-in 2 (1 arm) followed by DBDD Parallel Group Maintenance Period (2 arms) followed by optional Open-label Extension Period (1 arm)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded Site Rater, Blinded Clinical Research Associates (CRAs), active drugs and matching placebos are identical in their appearances.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- ND0612 Group (Experimental): ND0612 continuous SC infusion + Active IR-LD/CD (grey capsules) + Placebo IR-LD/CD (white capsules). Randomized DBDD Maintenance Treatment for 12 weeks.
  Interventions: Combination Product: ND0612 Solution for SC infusion; Drug: Oral IR-LD/CD; Drug: Placebo for Oral IR-LD/CD
- IR-LD/CD Group (Active Comparator): Placebo for ND0612 continuous SC infusion + Placebo IR-LD/CD (grey capsules) + Active IR-LD/CD (white capsules). Randomized DBDD Maintenance Treatment for 12 weeks.
  Interventions: Combination Product: Placebo for SC infusion; Drug: Oral IR-LD/CD; Drug: Placebo for Oral IR-LD/CD
- Oral IR-LD/CD Adjustment (Other): Active IR-LD/CD (white capsules). Open-label Treatment in Run-in 1 for 4-6 weeks.
  Interventions: Drug: Oral IR-LD/CD
- ND0612 Conversion (Other): ND0612 continuous SC infusion + Active IR-LD/CD (grey capsules). Open-label Treatment in Run-in 2 for 4-6 weeks.
  Interventions: Combination Product: ND0612 Solution for SC infusion; Drug: Oral IR-LD/CD
- Open-Label Extension (Other): ND0612 continuous SC infusion + Standard of care LD/dopa-decarboxylase inhibitor. Open-label Treatment in Extension for up to 54 months.
  Interventions: Combination Product: ND0612 Solution for SC infusion

INTERVENTIONS:
Combination Product: ND0612 Solution for SC infusion — Levodopa/Carbidopa (LD/CD) solution administered SC via infusion pump
  Arms: ND0612 Conversion; ND0612 Group; Open-Label Extension
Combination Product: Placebo for SC infusion — Placebo solution administered SC via infusion pump
  Arms: IR-LD/CD Group
Drug: Oral IR-LD/CD — Encapsulated LD/CD 100mg/25mg
  Other Names: IR-LD/CD
  Arms: IR-LD/CD Group; ND0612 Conversion; ND0612 Group; Oral IR-LD/CD Adjustment
Drug: Placebo for Oral IR-LD/CD — Encapsulated Placebo for LD/CD 100mg/25mg
  Other Names: Placebo for IR-LD/CD
  Arms: IR-LD/CD Group; ND0612 Group

SUMMARY:
This is a multi-center, randomized, double-blind, double-dummy, active controlled clinical Study. Following a screening period, eligible subjects will be enrolled to an open-label oral IR-LD/CD adjustment period; then an open-label ND0612 conversion period; then after optimization periods subjects will be randomized to receive either ND0612 or its matching Placebo with IR-LD/CD.

Subjects can continue to an optional open-label extension period.

DETAILED DESCRIPTION:
This is a phase III multi-center, randomized, active-controlled, double-blind, double-dummy (DBDD), parallel group clinical trial, investigating the efficacy, safety, and tolerability of continuous subcutaneous (SC) ND0612 infusion in comparison to oral IR-LD/CD in subjects with Parkinson's disease (PD) experiencing motor fluctuations.

This study is comprised of 6 periods:

1. a Screening Period;
2. an open-label oral IR-LD/CD Adjustment Period;
3. an open-label ND0612 Conversion Period;
4. a randomized DBDD active-controlled Maintenance Period;
5. an optional open-label Treatment Extension; and
6. a Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, aged ≥30 years.
2. PD diagnosis consistent with the United Kingdom Brain Bank Criteria.
3. Modiﬁed Hoehn & Yahr score ≤3 during "ON" state.
4. Average of ≥2.5 hours of OFF time (≥2 hours "OFF" time every day) during waking hours as conﬁrmed by patient diary over 3 days.
5. Taking ≥4 levodopa doses/day (≥3 doses/day of extended release LD/dopa-decarboxylase inhibitor, e.g., Rytary®) at a total daily dose of ≥400mg.

Exclusion Criteria:

1. Atypical or secondary parkinsonism.
2. Severe disabling dyskinesias, based on Investigator's discretion.
3. Previous neurosurgery for PD.
4. Use of duodenal levodopa infusion (LCIG) or apomorphine infusion.
5. Use of the following medications: subcutaneous apomorphine injections, sublingual apomorphine, or inhaled levodopa within 4 weeks.
6. Previous participation in ND0612 studies.
7. History of signiﬁcant skin conditions or disorders.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The change in daily ON time without troublesome dyskinesia | Baseline to the end of DBDD Maintenance Period (12 weeks)
  ON time without troublesome dyskinesia is the sum of ON time without dyskinesia and ON time with non-troublesome dyskinesia per patient diary

SECONDARY OUTCOMES:
The change in daily OFF time | Baseline to the end of DBDD Maintenance Period (12 weeks)
  OFF time per patient diary

CONTACTS AND LOCATIONS:
Overall Officials: Alberto J Espay, MD, MSc, Principal Investigator — University of Cincinnati OH, USA; Olivier Rascol, MD, PhD, Principal Investigator — Toulouse University Hospital, France
Locations (103):
- United States (38):
  - Xenoscience, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cedar- Sinai Medical Center Department of Neurology, Los Angeles, California
  - SC3 Research - Reseda, Reseda, California
  - University of California San Francisco, San Francisco, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Hartford Healthcare Chase Family Movement Disorders Center, Vernon, Connecticut
  - Visionary Investigators Network, Aventura, Florida
  - Parkinsons Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida Norman Fixel Institute for Neurological Diseases, Gainesville, Florida
  - Neurology Associates PA, Maitland, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Neurology One, Winter Park, Florida
  - Emory University - Brain Health Center, Atlanta, Georgia
  - NeuroStudies, Decatur, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Unity Point Health, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Neurology and Movement Disorder, Lexington, Kentucky
  - Oschner Medical Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - QUEST Research Institute, Farmington Hills, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai Medical center Movement Disorders Center, New York, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - Abington Neurological Associates LTD., Willow Grove, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Neurology Consultants of Dallas, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin Madison, Madison, Wisconsin
- Medical University Innsbruck, Innsbruck, Austria
- CHU de Tivoli, La Louvière, Belgium
- Czechia (2):
  - Neurologicka klinika Fakutni nemocnice sv. Anny v Brne, Brno
  - Axon Clinical s.r.o., Prague
- France (6):
  - Hopital Neurologique, Bron
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU Nantes-Hopital Laennec, Nantes
  - CHU de Nice Hpital Pasteur, Nice
  - Chu Caremeau, Nîmes
  - Hopital Purpan, Toulouse
- University of Pecs, Clinical Center, Pécs, Hungary
- Israel (6):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Ein Kerem, Jerusalem
  - Galilee Medical center- Nahariya, Nahariya
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Casa di Cura Villa Margherita, Arcugnano
  - Centro Ricerca Parkinson San Raffaele Cassino, Cassino
  - University Chieti CeSI MET Clinical research center-CRC, Chieti
  - Ospedale di Grosseto, Azienda USL Toscana Sud Est, Grosseto
  - Istituto Clinico Humanitas - IRCCS, Milan
  - AOU University of Campania "Luigi Vanvitelli", Naples
  - IRCCS Fondazione C. Mondino, Pavia
  - IRCCS San Raffaele Pisana, Roma
  - Policlinico Tor Vergata - UOSD Parkinson, Rome
  - IRCCS Santa Lucia Foundation, Rome
- University of Amsterdam, Amsterdam, Netherlands
- Poland (4):
  - Krakowska Akademia Neurologii Sp. z o. o, Krakow
  - NeuroKlinika Gabinet Lekarski Prof. Andrzej Bogucki, Lodz
  - Neuro-Care SP z o. o., Siemianowice Śląskie
  - Oddział Neurologii ul. L. Kondratowicza 8, Warsaw
- Portugal (2):
  - Hospital Braga, Braga
  - CNS - Campus Neurologico Senior, Torres Vedras
- Russia (5):
  - Kazan State Medical University, Kazan'
  - Federal Siberian Scientic Clinical Center of FMBA, Krasnoyarsk
  - Novosibirsk regional specialized scientific-practical neurological center on the basis City Clinical Hospital 34, Novosibirsk
  - The first Saint-Petersburg State Medical University named after IP Pavlov, Saint Petersburg
  - Siberian State Medical University, Tomsk
- Slovakia (2):
  - Nemocnica akad. L. Derera, Bratislava
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
- Spain (14):
  - Hospital Universitario central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Elche, Edificio principal, Alicante
  - Hospital Universitari de la Vall d'Hebron, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari General de Catalunya, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Infanta Sofia, Madrid
  - Hospital Universitario Virgen del Rocío, Laboratorio 104., Seville
  - Hospital Universitario y Politcnico de La Fe, Valencia
- Ukraine (5):
  - Clinic "Dopomoga Plus", Kyiv
  - Institute of Gerontolgoy - Parkinsons disease Treatment Centre, Kyiv
  - Ukrainian Medical Stomatological Academy based on Poltava Regional Clinical Hospital n.a. M.V.Skliphosovskyy, Poltava
  - Vinnytsia O.I. Yushchenko Regional Psychoneurology Hospital, Vinnytsia
  - Municipal Non-commercial Institution '' City hospital #9" of Zaporizhzhya City Council, Zaporizhzhya
- United Kingdom (5):
  - King's College hospital, London
  - St Georges University Hospital, London
  - Directorate of Medicine & Integrated Care, Imperial College Healthcare NHS Trust, London
  - Clinical Ageing research Unit, Newcastle
  - University Hospitals Plymouth NHS Trust, Plymouth

REFERENCES:
- [Derived] Espay AJ, Stocchi F, Pahwa R, Albanese A, Ellenbogen A, Ferreira JJ, Giladi N, Gurevich T, Hassin-Baer S, Hernandez-Vara J, Isaacson SH, Kieburtz K, LeWitt PA, Lopez-Manzanares L, Olanow CW, Poewe W, Sarva H, Yardeni T, Adar L, Salin L, Lopes N, Sasson N, Case R, Rascol O; BouNDless Study Group. Safety and efficacy of continuous subcutaneous levodopa-carbidopa infusion (ND0612) for Parkinson's disease with motor fluctuations (BouNDless): a phase 3, randomised, double-blind, double-dummy, multicentre trial. Lancet Neurol. 2024 May;23(5):465-476. doi: 10.1016/S1474-4422(24)00052-8. Epub 2024 Mar 15. PMID 38499015
- See also: European Union Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2018-004156-37/PT